CLINICAL TRIAL: NCT00494585
Title: Evaluation of CEP-701, an Orally Available JAK2 Tyrosine Kinase Inhibitor, as a Therapy for Patients With Myelofibrosis
Brief Title: CEP-701 for PH-negative Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0070; CS-2007-20040
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Results first posted 2011-05-04 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Leukemia; Myelofibrosis
Keywords: CEP-701; Leukemia; Myelofibrosis; MF; JAK2; Tyrosine Kinase Inhibitor; Lestaurtinib; Chronic Idiopathic Myelofibrosis; CIMF
MeSH Terms: conditions — Leukemia; Primary Myelofibrosis | interventions — lestaurtinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CEP-701 (Experimental): 80 mg orally twice a day for 30 days
  Interventions: Drug: CEP-701

INTERVENTIONS:
Drug: CEP-701 — 80 mg orally twice a day for 30 days
  Other Names: lestaurtinib

SUMMARY:
The goal of this clinical research study is to find out if CEP-701 can help control myelofibrosis (MF). The safety of CEP-701 will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

CEP-701 is designed to help prevent a certain type of molecule (called a mutated JAK2 receptor) that is found on myelofibrosis cells from sending continuous chemical signals that lead to the growth of cancer cells.

Study Treatment:

If you are found to be eligible to take part in this study, you will take CEP-701 by mouth (in liquid form) 2 times a day (once in the morning and once in the evening) every day in 30-day repeating cycles. You should take each dose about 12 hours apart.

The study doctor or nurse will teach you and/or a caregiver or family member how to prepare each dose of the study drug, as well as how much should be taken each time. At each study visit, you will be supplied with enough syringes, dosing cups, and study drug to last until your next study visit. For each dose, you will use the syringe to draw the proper amount of CEP-701. You will add the entire contents of the syringe to an approved juice in 1 of the provided dosing cups. You should also drink an additional dosing cup of juice after taking the drug dose. The following juices (100% juice only) are approved for use with CEP-701: grape, pineapple, apple, V8 vegetable juice, and orange juice.

The study drug mixture may be stored (in an areas that are protected from light, such as in a cabinet) for up to 1 hour at room temperature and up to 8 hours refrigerated (at about 35°F to 45 °F). If you miss a dose, you should not take another dose until your next scheduled dose.

Study Visits:

You will initially have study visits at M. D. Anderson once a month. You will need to return monthly for 6 months, then every 3 months if there are no side effects during the previous 3 cycles. After 2 years of therapy, your visits can be extended to every 6 months. After 6 cycles you may have either a study visit or a phone call from a member of study staff. If you have a phone call, you will be asked how you are feeling, if you have experienced any side effects since your last visit, and your blood tests will be reviewed with you. During most study visits, you will have the following tests:

* You will have a physical exam.
* You will be asked how you are feeling and about any side effects you may have experienced since your last visit.
* You will have blood (about 2 tablespoons) drawn to check your kidney and liver function and blood cell count. This will be done every 2 weeks up to 3 months, then every 1-2 months.
* You will have a bone marrow/aspirate once every 3-6 months to see if you are responding to treatment. After 2 years of therapy, this can be extended to every 12 months.

Length of Study:

You will continue on this study for at least 6 months to allow time for response. If you do respond to study treatment, you may continue to receive cycles for up to 5 years.

If you do not respond to study treatment within 6 months, if the disease gets worse, if intolerable side effects occur, if you have an illness that keeps you from taking the study drug, or your doctor thinks it is in your best interest to stop taking part in this study, you will be taken off this study.

This is an investigational study. CEP-701 is not Food and Drug Administration (FDA) approved or commercially available. At this time, it is being used for research purposes only in this study. Up to 41 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Idiopathic Myelofibrosis (CIMF) requiring therapy, including those 1) previously treated by CIMF-directed therapy and relapsed, intolerant, or refractory to therapy; or 2) if newly diagnosed then with intermediate or high risk according to Lille scoring system (adverse prognostic factors are: Hb < 10 g/dl, WBC < 4 or > 30 x 10^9/L; risk group: 0 = low, 1 = intermediate, 2 = high), or with symptomatic spleen that is >/= 10cm below costal margin. However, patients with asymptomatic intermediate risk disease are not eligible.
* JAK2 mutation positive test
* Age of at least 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate liver and renal function: total bilirubin </=2.0 mg/dL, alanine aminotransferase (ALT or SGPT) </=2.0 x institutional upper limit of normal (ULN), and creatinine </=2.0 mg/dl
* Patients must be at least 2 weeks from prior chemotherapy, biological therapy, radiation therapy, major surgery, or other investigational anticancer therapy that is considered MF-directed, and have recovered from prior toxicities to Grade 0-1. Concurrent therapy with supportive care medications (hydroxyurea, anagrelide) is allowed during the study.
* All men of reproductive potential and women of child-bearing potential (WOCBP) must agree to practice effective contraception (iud, birth control pill, latex condoms, diaphragm) during the entire study period and for one month after the study ends, unless documentation of infertility exists. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. WOCBP are women who are not menopausal for 12 months or no previous surgical sterilization."
* Ability to understand and willingness to sign the informed consent form
* Not willing to undergo, not a candidate for, or not having a donor for, a bone marrow transplant

Exclusion Criteria:

* Pregnant or nursing women, due to the unknown effects of therapy on the developing fetus or newborn infant.
* Patients diagnosed with another malignancy - unless following curative intent therapy the patient has been disease free for at least 3 years. Patients with early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia (CIN) are eligible for this study
* Any condition, including serious medical condition, laboratory abnormality, or psychiatric illness, which places the subject at unacceptable risk as judged by the Principal Investigator, if he/she was to participate in the study
* Known positive for Human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C
* Presence of any gastrointestinal condition or concomitant medication use (e.g. coumadin) that would render a patient at high risk for gastrointestinal bleeding as judged by treating physician
* History of any upper or lower gastrointestinal bleeding in the 6 months prior to enrollment
* Elevated international normalized ratio (INR) or Partial thromboplastin time (PTT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Santos FP, Kantarjian HM, Jain N, Manshouri T, Thomas DA, Garcia-Manero G, Kennedy D, Estrov Z, Cortes J, Verstovsek S. Phase 2 study of CEP-701, an orally available JAK2 inhibitor, in patients with primary or post-polycythemia vera/essential thrombocythemia myelofibrosis. Blood. 2010 Feb 11;115(6):1131-6. doi: 10.1182/blood-2009-10-246363. Epub 2009 Dec 11. PMID 20008298
- See also: M.D. Anderson's website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 6/28/2007 through 10/25/2007. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 27 participants registered, 5 participants were ineligible to participate.
Groups:
- CEP-701: 80 mg orally twice daily for 30 days
Period: Overall Study
Arm/Group | CEP-701
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CEP-701
Number analyzed (Participants) | 22
Age Continuous [Median (Full Range); unit: years] | 61 [38 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response = Complete Response, absence sign/symptoms of disease (without use of growth factors, hydroxyurea, anagrelide, or transfusions for > 1 month); Partial Response, absence of progressive disease (PD), and improvement in 2+ parameters (if abnormal): Absolute neutrophil count (ANC), hemoglobin, platelets, transfusions, splenomegaly, or bone marrow blasts; Clinical Improvement, absence of PD, and improvement in 1 parameter: ANC, hemoglobin, platelets, transfusions, splenomegaly, or bone marrow blasts). [International Working Group on Myelofibrosis Research and Treatment]
Time Frame: Response assessed after each 3 cycles (cycle = 30 days)
Population: Intention to treat.
Measure: Number; unit: Participants
Arm/Group | CEP-701
Number analyzed (Participants) | 22
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Clinical Improvement (CI) | 6

ADVERSE EVENTS:
Time Frame: 3 years 10 months
Arm/Group | CEP-701
Serious Adverse Events (participants affected / at risk) | 7/22
Other Adverse Events (participants affected / at risk) | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEP-701 (N=22)
Hematoma (Blood and lymphatic system disorders) | 1 (1) — Due to an accident
Debridement surgery with VAC placement (General disorders) | 1 (1) — After an accidental fall
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) — Due to a fall
Death (General disorders) | 4 (4) — Disease Progression
Chronic Interstitial Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEP-701 (N=22)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 16 (16)
Nausea (Gastrointestinal disorders) | 11 (11)
Headache (Nervous system disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 6 (6)
Flatulence (Gastrointestinal disorders) | 5 (5)
Heartburn (Gastrointestinal disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 3 (3)
Peripheral Neuropathy (Nervous system disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 6 (6)
Elevated alanine aminotransferase (Hepatobiliary disorders) | 6 (6)
Elevated alkaline phosphatase (Hepatobiliary disorders) | 2 (2)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes